CLINICAL TRIAL: NCT04624087
Title: The Effect of Go/No-Go Training Dosage on Weight Loss, Food Evaluation, and Disinhibition in Overweight and Obese Individuals: A Randomized Controlled Trial
Brief Title: Go/No-Go Intervention for Weight Loss
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Minnesota (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 00010522
Record Dates: First submitted 2020-10-13; First posted 2020-11-10 (Actual); Last update posted 2022-03-21 (Actual); Status verified 2022-03

CONDITIONS: Overweight and Obesity
MeSH Terms: conditions — Overweight; Obesity

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- High Dose (Experimental): Participants will perform the food-specific computerized go/no-go training four times per week for 4 weeks.
  Interventions: Behavioral: food-specific go/no-go computerized training
- Low Dose (Experimental): Participants will perform the food-specific computerized go/no-go training one time per week for 4 weeks.
  Interventions: Behavioral: food-specific go/no-go computerized training
- Active Control (Active Comparator): Participants will perform the generalized, nonfood-specific computerized go/no-go training one time per week for 4 weeks.
  Interventions: Behavioral: nonfood-specific go/no-go computerized training

INTERVENTIONS:
Behavioral: food-specific go/no-go computerized training — Participants will perform the computerized food specific go/no-go training a designated number of times over a four week duration (frequency varies by group). Each training session will last approximately 10 minutes and occur on different days of the week.
  Arms: High Dose; Low Dose
Behavioral: nonfood-specific go/no-go computerized training — Participants will perform the computerized general go/no-go training 1 time per week over a four week duration. Each training session will last approximately 10 minutes and occur on different days of the week.
  Arms: Active Control

SUMMARY:
The purpose of this study is to assess the effect of a food-specific Go/No-Go (GNG) computerized training task on weight loss, food evaluation, and disinhibition in a population of overweight and obese individuals.

DETAILED DESCRIPTION:
Within the current obesogenic environment, the prevalence of overweight and obesity has dramatically increased over the past 40 years. As a result, approximately 40% of Americans attest to being on a diet, with most of these efforts being unsuccessful. Most weight loss diets rely on self-control and reflective thinking (e.g., making conscious food choices multiple times per day), despite the fact that responses to appetitive foods often occur through implicit (unconscious) processes. The proposed study is a randomized clinical trial for weight loss that targets these implicit processes through the use of a computerized, food-specific, go/no-go task. This task has previously resulted in reduced food consumption in laboratory settings, and small but significant weight loss in two brief intervention studies. The purpose of this study is to replicate one prior study and to compare different doses of the intervention. Participants will be assigned to one of three groups: high intensity, low intensity, or active control, and will be assessed on a number of variables pre- and post-intervention. Changes in body weight, food evaluation, frequency of self-reported food consumption, and eating disinhibition scores will be evaluated. It is hypothesized that individuals receiving the food-specific go/no-go training (high intensity and low intensity groups) will experience greater weight loss, decreased disinhibition with food, and reduced snacking of the targeted foods than those in the active control group. It is also hypothesized that the high intensity intervention will be more effective than the low intensity intervention across these variables. Moderators (e.g., dietary restraint, disinhibition) will also be explored throughout this study, along with the mechanism of devaluation of specific foods.

ELIGIBILITY:
Inclusion Criteria:

* Body Mass Index (BMI) ≥ 25
* Age ≥ 18
* Consume some of the determined "no-go" snack foods at least three times per week (assessed using a food frequency questionnaire)
* A desire to lose weight

Exclusion Criteria:

* Medical condition limiting dietary intake
* Medical condition directly affecting weight
* Current use of weight loss medication
* Actively enrolled in a formal weight loss program currently or within the past 6 months (e.g., Weight Watchers)
* History of bariatric surgery
* Currently pregnant
* Current smoker
* Smoking cessation within the past year

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 78 (Actual)
Dates: Start 2020-10-19 (Actual); Primary Completion 2021-11-01 (Actual); Study Completion 2021-11-01 (Actual)

PRIMARY OUTCOMES:
Change in body weight from baseline to post 4-week intervention, to 6-month follow-up | baseline, post 4-week intervention, 6-month follow-up
  Body weight will be measured by participant using personal or university scale. Participants will take a picture of their weight send it to the research team (Due to COVID-19 precautions, in person weighing is not possible).
Change in disinhibition scores from baseline to post 4-week intervention, to 6-month follow-up. | baseline, post 4-week intervention, 6-month follow-up
  This will be measured using the Disinhibition subscale of the Three Factor Eating Questionnaire; minimum value = 0; maximum value = 16; higher scores for this measure means worse outcomes
Change in frequency of food consumption from baseline to post 4-week intervention, to 6-month follow-up. | baseline, post 4-week intervention, 6-month follow-up
  This will be measured using a food frequency questionnaire assessing food intake over the previous month.

SECONDARY OUTCOMES:
Change in binge eating behaviors from baseline to post 4-week intervention, to 6-month follow-up. | baseline, post 4-week intervention, 6-month follow-up
  This will be measured using the binge eating questions of the Eating Disorder Examination Questionnaire; minimum value = 0; maximum value = unlimited; higher scores for this measure means worse outcomes
Change in liking of foods from baseline to post 4-week intervention, to 6-month | baseline, post 4-week intervention, 6-month follow-up
  This will be measured using a visual analog scale; minimum value = -100; maximum value = 100; higher scores for this measure on healthy foods means better outcomes, higher scores on this measure for unhealthy foods means worse outcomes
Change in automatic responses to healthy and unhealthy foods from baseline to post 4-week intervention, to 6-month | baseline, post 4-week intervention, 6-month follow-up
  This will be measured using an impulsive food choice test.

CONTACTS AND LOCATIONS:
Overall Officials: Lara LaCaille, PhD, Principal Investigator — University of Minnesota
Locations (1):
- University of Minnesota Duluth, Duluth, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No